CLINICAL TRIAL: NCT01160172
Title: A Partially Blind Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Staphylococcal 4-component Investigational Vaccine (GSK2392102A) in Healthy Adults
Brief Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Staphylococcal Investigational Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113949
Record Dates: First submitted 2010-07-01; First posted 2010-07-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Infections, Staphylococcal
Keywords: vaccine; young adults; Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (6):
- Group A (Experimental)
  Interventions: Biological: Staphylococcal investigational vaccine GSK2392103A
- Group B (Experimental)
  Interventions: Biological: Staphylococcal investigational vaccine GSK2392105A
- Group C (Experimental)
  Interventions: Biological: Staphylococcal investigational vaccine GSK2392106A
- Group D (Experimental)
  Interventions: Biological: Staphylococcal investigational vaccine GSK2392019A
- Group E (Placebo Comparator)
  Interventions: Drug: Saline placebo
- Group F (Placebo Comparator)
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Biological: Staphylococcal investigational vaccine GSK2392103A — intramuscular vaccination according to protocol schedule
  Arms: Group A
Biological: Staphylococcal investigational vaccine GSK2392105A — intramuscular vaccination according to protocol schedule
  Arms: Group B
Biological: Staphylococcal investigational vaccine GSK2392106A — intramuscular vaccination according to protocol schedule
  Arms: Group C
Biological: Staphylococcal investigational vaccine GSK2392019A — intramuscular vaccination according to protocol schedule
  Arms: Group D
Drug: Saline placebo — intramuscular vaccination according to protocol schedule
  Arms: Group E; Group F

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of several formulations of an investigational Staphylococcal vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female between 18 and 40 years of age, inclusive, at the time of first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history, clinical examination and laboratory assessment before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test at Screening, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* Any clinically significant acute or chronic, local or systemic infection, proven or suspected to be caused by Staphylococcus aureus and requiring antibiotic treatment, within the 6 months preceding the first vaccination.
* Previous administration of any investigational Staphylococcus aureus vaccine/antibodies.
* History of; or current bleeding or coagulation disorder.
* Known or suspected reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of; or current autoimmune or other immune-mediated disease.
* Administration or planned administration, of any vaccine not foreseen by the study protocol within 30 days of the first dose of vaccines up to 1 month after the last vaccine dose.
* Administration of immunoglobulins and/or any blood products within the last 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Any clinically relevant abnormal haematological or biochemical or urine laboratory values at screening.
* Any acute or chronic, clinically significant disease, as determined by physical examination or laboratory screening tests.
* Acute disease and/or fever at study entry.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of; or current alcoholism and/or drug abuse.
* Any other condition that the principal investigator judges may interfere with study findings.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2010-07-19 (Actual); Primary Completion 2012-08-23 (Actual); Study Completion 2012-08-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited local and general adverse events (AEs) in all subjects, in all vaccine groups. | During a 7-day (day 0-6) follow up period after each vaccine dose
Occurrence of unsolicited adverse events (AEs) in all subjects, in all vaccine groups. | During a 30-day (day 0-29) follow up period after each vaccine dose
Occurrence of any Serious Adverse events (SAE) in all subjects, in all vaccine groups. | From first vaccination (Day 0) to study conclusion (Day 540)
Occurrence of any adverse event (AE) of specific interest in all subjects, in all vaccine groups. | From first vaccination (Day 0) to study conclusion (Day 540)
Occurrence of haematological, biochemical or urinary laboratory abnormalities in all subjects, in all vaccine groups. | Prior to each vaccine dose
Occurrence of haematological, biochemical or urinary laboratory abnormalities in all subjects, in all vaccine groups. | 1 day after each vaccine dose
Occurrence of haematological, biochemical or urinary laboratory abnormalities in all subjects, in all vaccine groups. | 7 days after each vaccine dose
Occurrence of haematological, biochemical or urinary laboratory abnormalities in all subjects, in all vaccine groups. | 29/30 days after each vaccine dose
Occurrence of haematological, biochemical or urinary laboratory abnormalities in all subjects, in all vaccine groups. | 6 months after the last vaccine dose
Occurrence of haematological, biochemical or urinary laboratory abnormalities in all subjects, in all vaccine groups. | 12 months after the last vaccine dose

SECONDARY OUTCOMES:
Immune response to components of the Staphylococcal vaccine formulations in all subjects, in all vaccine groups. | Prior to each vaccine dose, 1, 7 and 29/30 days after each vaccine dose, and 6 and 12 months after the last vaccine dose.
Colonisation with Staphylococcus aureus in all subjects, in all vaccine groups. | At Screening (pre-Day 0) and at Days 0, 30, 60, 180, 210 and 540.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, La Louvière, Belgium

REFERENCES:
- [Derived] Levy J, Licini L, Haelterman E, Moris P, Lestrate P, Damaso S, Van Belle P, Boutriau D. Safety and immunogenicity of an investigational 4-component Staphylococcus aureus vaccine with or without AS03B adjuvant: Results of a randomized phase I trial. Hum Vaccin Immunother. 2015;11(3):620-31. doi: 10.1080/21645515.2015.1011021. PMID 25715157
- See also: Results for study 113949 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/113949?search=study&b%22b''%22#rs